CLINICAL TRIAL: NCT04315701
Title: Evaluating the PD-1 Checkpoint Inhibitor, Cemiplimab, as Neoadjuvant Therapy in High Risk Localized, Locally Recurrent, and Regionally Advanced Cutaneous Squamous Cell Carcinoma: A Phase II Pilot Study
Brief Title: A PD-1 Checkpoint Inhibitor (Cemiplimab) for High-Risk Localized, Locally Recurrent, or Regionally Advanced Skin Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14SK-19-1; NCI-2020-01247 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14SK-19-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Skin Squamous Cell Carcinoma; Resectable Skin Squamous Cell Carcinoma; Stage I Skin Cancer; Stage II Skin Cancer; Stage III Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cemiplimab, surgical resection) (Experimental): Patients receive cemiplimab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles (or up to 4 cycles for patients whose disease is unresectable after 3 cycles) in the absence of disease progression or unacceptable toxicity. Within 6 weeks of last dose of therapy, patients with potentially resectable tumors undergo surgical resection.
  Interventions: Biological: Cemiplimab; Procedure: Resection

INTERVENTIONS:
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN2810
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase II trial studies how well cemiplimab before surgery works in treating patients with skin cancer that is high-risk and has not spread to other parts of the body (localized), has come back locally (locally recurrent), or has spread regionally (regionally advanced), and can be removed by surgery (resectable). Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the pathological partial response (PPR) rate in patients with potentially resectable cutaneous squamous cell carcinoma (CSCC) treated with neoadjuvant cemiplimab.

SECONDARY OBJECTIVES:

I. To estimate the pathological complete response rate (PCR). II. To estimate the Response Evaluation Criteria in Solid Tumors (RECIST) (version [v]1.1) 9 week objective response rate (ORR).

III. To estimate the RECIST (v1.1) 12 month progression free (PFS). IV. To assess the toxicity among patients with CSCC treated with neoadjuvant cemiplimab.

EXPLORATORY OBJECTIVES:

I. To evaluate tumor mutational burden (TMB) and correlate with response to PD-1 blockade therapy.

II. To evaluate PD-L1 expression on CSCC tumor cells and correlate with response to PD-1 blockade.

III. To evaluate CD8+ T cell infiltration into CSCC tumors and correlate with response to PD-1 blockade.

IV. To assess other adaptive immune resistance mechanisms in CSCC tumors.

OUTLINE:

Patients receive cemiplimab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles (or up to 4 cycles for patients whose disease is unresectable after 3 cycles) in the absence of disease progression or unacceptable toxicity. Within 6 weeks of last dose of therapy, patients with potentially resectable tumors undergo surgical resection.

After completion of study treatment, patients are followed up every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, cutaneous squamous cell carcinoma
* Patients must have disease that is deemed potentially resectable, at the time of the start of study, by the treating investigator. The decision to perform surgery on patients must be based on good clinical judgment. Eligible patients for surgical resection must have disease that, in the judgment of the surgeon, is deemed potentially resectable, resulting in free surgical margins
* Patients must have measurable disease
* Patients must have disease that is considered either: (1) high-risk localized CSCC, (2) locally recurrent CSCC, or (3) regionally advanced CSCC. The criteria specific to each of these populations is listed below

  * For patients with high-risk localized CSCC, at least two of the following clinical or pathologic high-risk features must be present to be eligible:

    * Clinical risk factors

      * Any tumor size > 2.0 cm in diameter
      * Tumors > 1.0 cm in high risk locations, including "mask areas" (central face, eyelids, eyebrow, nose, lips [cutaneous], periorbital, chin, mandible, preauricular and postauricular skin/sulci, genitalia, hands, feet, cheek, forehead, scalp, neck and pretibial)
      * Any rapidly growing and/or symptomatic tumor
    * Pathologic risk factors

      * Poorly differentiated histology
      * Depth > 6 mm in thickness
      * Acantholytic / adenoid, adenosquamous, desmoplastic, or metaplastic / carcinosarcomatous histologic subtypes
      * Invasion beyond subcutaneous fat
      * Perineural, lymphatic, or vascular involvement
  * Patients with locally recurrent CSCC, that failed prior surgery, radiation or systemic therapy, are eligible, as long as they have measurable disease and are deemed potentially resectable by the treating investigator
  * Patients with regionally advanced CSCC, including in-transit, cutaneous, subcutaneous or lymph node metastases are eligible, as long as they have measurable disease and are deemed potentially resectable by the treating investigator
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count >= 1,000 /mcL
* Absolute lymphocyte count >= 500 / mcL
* Hemoglobin >= 8.0 g/dL
* Platelets >= 75,000/mcl
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT]) =< 3 x institutional upper limit of normal
* Creatinine =< 1.8 mg/dl
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Ability to understand and the willingness to sign a written informed consent and comply with surgical resection at end of study and other study-related procedures

Exclusion Criteria:

* Metastatic disease that is unresectable. Patients with visceral metastases are not eligible. Regionally advanced disease, including in-transit, cutaneous, subcutaneous, or nodal metastases are allowed, if deemed potentially resectable by the investigator
* Prior treatment with cemiplimab or any other agent that blocks the PD-1 or PD-L1 pathway
* Prior treatment with other immune modulating agents within fewer than 4 weeks, prior to the first dose of cemiplimab. Examples of immune modulating agents include blockers of CTLA-4, 4-1BB, OX-40, therapeutic vaccines, or cytokine therapies
* Patients must not be receiving other concomitant biologic therapy, hormonal therapy, chemotherapy, other anti-cancer therapy or any other investigational agents while on this protocol
* Radiation therapy, non-cytotoxic agents or investigational agents in the 4 weeks prior to registration
* Immunosuppressive systemic corticosteroids equivalent to prednisone 10 mg or greater in the 14 days prior to the first dose of cemiplimab
* Any major surgery within 14 days prior to the first dose of cemiplimab. Patients must have recovered from any major complications before registration
* Active autoimmune disease requiring systemic treatment in the past 2 years (i.e. use of disease modifying agents or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment
* History of other prior malignancy in the last five years, with the exception of: adequately treated non-melanoma skin cancers (including multiple primary skin cancers), adequately treated in situ cancer, and other local tumors considered cured by local treatment (including melanoma)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cemiplimab or any other PD-1 or PD-L1 inhibitor
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness / social situations that would limit compliance with study requirements
* Positive pregnancy test, active pregnancy or nursing / breast-feeding, due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
* History solid organ or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2027-06-17 (Estimated)

PRIMARY OUTCOMES:
Confirmed pathologic partial response | Up to 24 months after completion of study treatment
  Defined by presence of < 50% malignant cells. Descriptive statistics will be used to summarize the measurements.

SECONDARY OUTCOMES:
Pathologic complete response rate | Up to 24 months after completion of study treatment
  Descriptive statistics will be used to summarize the measurements.
Objective response rate | At 9 weeks
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Descriptive statistics will be used to summarize the measurements.
Progression-free survival | From start of treatment to time of progression or death whichever comes first, assessed at 12 months
  Measured by RECIST v1.1. Descriptive statistics will be used to summarize the measurements.
Incidence of toxicities | Up to 24 months after completion of study treatment
  All toxicities will be summarized and graded according to maximum grade by Common Terminology Criteria for Adverse Events v4. Descriptive statistics will be used to summarize the measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Gino K In, MD, Principal Investigator — University of Southern California
Locations (5):
- United States (5):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Nebraska, Omaha, Nebraska